CLINICAL TRIAL: NCT00709579
Title: Physiopathological Study and Pharmacological Modulation of Cutaneous Atrophy's Markers Induced by Glucocorticoids
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Collaborators: University Paul Sabatier of Toulouse (Other); University Hospital, Geneva (Other); Centre Européen de Recherche sur la Peau, (Unknown); Pierre Fabre BIOMETRIE (Unknown)
Responsible Party: Anne-Marie SCHMITT, Pierre Fabre Dermo Cosmetique
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MODULCORTICOATROPHIE; 2007-A00675-48
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Cortico Atrophy
Keywords: Patients needing an oral corticotherapy; Patients needing a topical corticotherapy; Corticotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RV3391A (Active Comparator)
  Interventions: Drug: RV3391A

INTERVENTIONS:
Drug: RV3391A — A standardized quantity of each product will be applied on the evening on anterior side of forearm. The side of application will be randomized.
  Arms: RV3391A
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
Methodology :Phase III study, single centre, double blind, versus excipient, randomised, controlateral design.

Selection of the patients :Number of subjects required 60 :

* 30 patients needing an oral corticotherapy
* 30 patients needing a topical corticotherapy

DETAILED DESCRIPTION:
Study conduct

Two steps for each patient:

1. the first step lasting 3 months : assessment of changes in mechanisms involved in ACIC with the RV3391A cream (M0 à M3). At the beginning of the corticotherapy, each patient will apply RV3391A on anterior side of a forearm and the placebo on the other side (randomised) for 3 months.

   Clinical exam and objective measurements will be realised.

   This step will allow us to describe and compare the evolution of cutaneous atrophy's markers produced by glucocorticoïds markers between M0 and M3:
   * between topical and oral corticotherapy
   * between RV3391A and the placebo.
2. the second step, the cohort follow-up, leading off the end of the first step (M3 à M24) The period of the second step will depend on the progression of patient's disease and on the period of his medical follow-up. This period may lasting until the 24th month after the inclusion in the study.

The patients will not apply RV3391A and the placebo anymore. They will be followed-up in the CHU.Assessments of the cutaneous atrophy's markers produced by glucocorticoïds will be realised at M6, M12, M18 and M24 with non invasive methods (clinical scoring, imaging, extensometry) to exactly describe on a long-term period the evolution of the ACIC. The assessments on forearm having received the placebo will allow us to know natural history of skin atrophy induced by corticotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing an oral corticotherapy:

  * aged over 50 years
  * first corticotherapy over 0.5 mg/kg/day
  * expectable period with a corticotherapy over 10 mg/day more than 3 months
  * having signed a written informed consent form
  * registered with a social security or health insurance system
* Patients needing a topical corticotherapy:

  * aged over 50 years
  * topical corticotherapy with a high or very high potency corticoid over 10 g/day
  * expectable period with a topical corticotherapy more than 3 months
  * having signed a written informed consent form
  * registered with a social security or health insurance system

Exclusion Criteria:

* Oral or topical corticotherapy within the last 3 months
* Cutaneous inflammation on the anterior side of the forearm
* Medical history of psychosis induced by corticotherapy
* Medical history of allergy to RV3391A product its and excipients.
* Medical history of allergy to mineral cream Avene SPF50 excipients.
* Medical history of allergy to latex, surgical tape, chlorhexidine, lidocaine or xylocaine
* Clotting disorder or anticoagulant intake
* Healing disorder
* Women who are not post-menopausal women
* Substitutive estrogenotherapy for less than 6 months
* Impossibility to be registered in the Volunteers National Register
* Inability to comply with requirements of the clinical monitoring program,
* Inability to personally sign the informed consent form
* Is deprived of his freedom by an administrative or judicial decision; or who is under guardianship or protective custody

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
20 Mhz echography : Dermal Thickness | M0 versus M3

SECONDARY OUTCOMES:
20 Mhz echography : Dermal Thickness | M0 versus M6, M12, M18, M24
Optical Coherent Tomography : Epidermal Thickness | M0, M1, M3, M6, M12, M18, M24
Frosch Score | M0, M1, M3, M6, M12, M18, M24
Cutometry: assessment of the skin mechanical properties | M0, M1, M3, M6, M12, M18, M24
Histology: study of skin layers and assessment of collagen and other proteins. | M0, M3
Immunohistology and molecular biology: assessment of CD44, HB-EGF and erbB1, cutaneous cytokines, filaggrin, corneodesmosin and involucrin. | M0, M3
Peeling with an adhesive tape: sample of superficial epidermis layers and assessment by biochemical and immunodetection methods of anti-desmoglein, anti-kallikrein 7 and anti-corneodesmosin antibodies | M0, M3,

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Sailler, Professor, Principal Investigator — Centre Hospitalier Universitaire; Anne-Marie Schmitt, Doctor, Study Director — Pierre Fabre Dermo Cosmetique; Carle Paul, Professor, Study Director — Centre Hospitalier Universitaire
Locations (1):
- Centre Hopitalier Universitaire de Toulouse, Toulouse, France